CLINICAL TRIAL: NCT06769477
Title: The Effect of Training With Motivational Interviewing Based on Health Belief Model on Diabetes Self-Management, Health Fatalism and Metabolic Parameters in Individuals With Type 2 Diabetes: A Randomized Controlled Experimental Study
Brief Title: The Effect of Education Given to Type 2 Diabetics on Diabetes Self-management, Health Fatalism and Metabolic Parameters
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Gülşen Altuntas Çalım, health services teacher in the ministry of national education, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AU-SBF-GAÇ-01
Record Dates: First submitted 2025-01-07; First posted 2025-01-10 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Type 2 Diabetes; Type 2 Diabetes Patients
Keywords: health belief model; motivational interview; self-management; health fatalism; type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: the experimental group will be trained with motivational technique. the control group will not receive any intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group receiving diabetes education with motivational interviewing technique (Active Comparator): Patient Introduction Form, Type 2 DM Self-Management Scale (SMS) and Health Fatalism Scale will be applied to the experimental group before the training. then, diabetes education will be given to the individuals in the experimental group one day a week with the motivational interviewing technique based on the health belief model. 8 weeks of training will be given in total and then 4 weeks of informative reminder sms will be sent about diabetes education. After the training is over, Patient Introduction Form, Type 2 DM Self-Management Scale (SMS) and Health Fatalism Scale will be applied.
  Interventions: Other: Experimental Group
- group with no intervention (No Intervention): The control group will be administered the Patient Introduction Form, Type 2 DM Self-Management Scale (SMS) and Health Fatalism Scale at the first encounter. After 3 months, the Patient Introduction Form, Type 2 DM Self-Management Scale (SMS) and Health Fatalism Scale will be applied again. No application will be made to the control group.

INTERVENTIONS:
Other: Experimental Group — individuals will receive diabetes education with motivational interviewing technique based on health belief model
  Arms: group receiving diabetes education with motivational interviewing technique

SUMMARY:
This study aims to examine the effects on diabetes self-management, health fatalism and metabolic parameters of individuals with type 2 diabetes. The study will be conducted in a health institution between February 2025 and May 2025 and participants will be assigned to experimental and control groups by simple random sampling method. The experimental group will be trained with motivational interviewing techniques based on the health belief model for 8 weeks, followed by sending reminder SMS for 4 weeks. The control group will receive no intervention. The study is expected to improve the self-care behaviors of individuals with diabetes by creating positive effects on diabetes management and health fatalism.

DETAILED DESCRIPTION:
This study aims to determine the effect of education given with motivational interviewing technique structured according to the health belief model on diabetes self-management, health fatalism and metabolic parameters in individuals with type 2 diabetes. The research will be conducted in a pre-test and post-test randomized controlled experimental design.The population of the study will consist of individuals with type 2 diabetes who are registered in a health institution between February 2025 and May 2025 and who meet the research criteria. The sample determined by power analysis will consist of a total of 66 patients, 33 in the experimental group and 33 in the control group. Patient Introduction Form, Type 2 DM Self-Management Scale (SMS) and Health Fatalism Scale will be used to collect data from the experimental and control groups for pre-test and post-test. Weight, height, waist circumference and body mass index of the individuals will be measured by the researcher and HbA1c values of the last one month will be recorded. The experimental group will be given diabetes education with motivational interviewing technique structured according to the health belief model in line with the literature.Brochures and powerpoint presentations will be prepared as training materials. Trainings will be held in the training room on the days and times determined with the patients in 8 sessions lasting 30-40 minutes. At the end of the training, an SMS message will be sent once a week for four weeks. At the end of each visit, the next visit will be scheduled. Trainings will be conducted face-to-face by the researcher. The control group will not receive any training. After the completion of the trainings, a post-test will be administered to both the experimental and control groups. In the evaluation of the data; numbers, percentages, standard deviation, mean, minimum and maximum values, Chi-square, Fisher-Freeman-Halton Exact Test, Paired Samples t-test and Independent Samples t-test will be used.

ELIGIBILITY:
Inclusion Criteria:

* Having type 2 diabetes for at least 6 months
* To be over 18 years old
* Have sufficient communication skills to answer verbal and written questions and fulfill instructions
* Becoming literate
* No physical, cognitive or mental impairment in answering the questions
* Willingness to participate in research.

Exclusion Criteria:

* Under 18 years of age
* Being hospitalized in inpatient treatment institutions due to DM or DM complications during the research process
* The emergence of any health problem that prevents the person from continuing the research
* Do not leave the study voluntarily.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Type 2 DM Self-Management Scale (SMS) | three months
  The scale assesses self-management It has 3 sub-dimensions.These dimensions consist of 11 questions consisting of "Healthy Lifestyle Behaviors" dimension, consisting of 4 questions "Health Services Utilization" dimension and "Blood Sugar Management" dimension. Scoring: Always 5, Often 4, Sometimes 3, Rarely 2, Never 1.
  (-Healthy Lifestyle Subdimension= HLBD-1+ HLBD-2+ HLBD-3+ HLBD-4+ HLBD-5+ HLBD-6+ HLBD-7+ SYBD-8+ SYBD-9+ SYBD-10+ SYBD-11.) (-Blood Glucose Management Subscale= BSM-1+ BSM-2+ BSM-3+ BSM-4) (-Health Services Utilization Subdimension= SHK-1+ SHK-2+ SHK-3+ SHK-4) (-Diabetes Self-Management Scale score=SMDI Subdimension+CSM Subdimension +SCC Subdimension.) There are no reverse items in the scale. High scores indicate good self-management, low scores indicate and poor self-management. The minimum score that can be obtained from the Type 2 self-management scale is 19 and the maximum score is 95.

SECONDARY OUTCOMES:
Health Fatalism Scale | three months
  The scale consists of one sub-dimension and 17 items. The scale is a Likert-type scale answered as ''strongly disagree'', ''disagree'', ''undecided'', ''agree'', ''strongly agree''. The minimum score obtained from the Health Fatalism Scale is 17 and the maximum score is 85. Cronbach α Coefficient of the scale is 0.91.An increase in the score on the scale indicates an increase in fatalism.

CONTACTS AND LOCATIONS:
Locations (1):
- Manavgat and Aksu Family Health Center, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No